CLINICAL TRIAL: NCT06435312
Title: An Open-Label Extension Study to Evaluate the Long-Term Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Activity of Zilucoplan in Pediatric Study Participants With Acetylcholine Receptor Antibody Positive Generalized Myasthenia Gravis
Brief Title: An Open-label Extension Study to Evaluate Subcutaneous Zilucoplan in Pediatric Participants With Generalized Myasthenia Gravis
Acronym: ziMyG+
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MG0015; 2022-502073-42 (Registry Identifier: EU Clinical Trials); U1111-1290-3806 (Other: World Health Organization (WHO))
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Generalized Myasthenia Gravis
Keywords: generalized Myasthenia Gravis; gMG; RA101495; Zilucoplan; pediatric; MG0015
MeSH Terms: conditions — Myasthenia Gravis | interventions — zilucoplan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Zilucoplan Arm (Experimental): Study participants will receive Zilucoplan at a pre-defined dose based on their weight.
  Interventions: Drug: Zilucoplan

INTERVENTIONS:
Drug: Zilucoplan — Zilucoplan will be administered subcutaneously to pediatric study participants
  Other Names: RA101495

SUMMARY:
The purpose of this study is to assess the long-term safety and tolerability of an additional 52 weeks of Zilucoplan treatment administered by subcutaneous injection once daily in pediatric study participants

ELIGIBILITY:
Inclusion Criteria:

United States of America (USA) specific inclusion criterion:

- Participant must be ≥ 12 years of age at the time of signing the Informed Consent/Assent according to local regulation.

Rest of World (ROW) specific inclusion criterion:

- Participant must be ≥ 2 years of age at the time of signing the Informed Consent/Assent according to local regulation.

Global specific inclusion criteria:

* Participant has completed the MG0014 according to the protocol, and further treatment with zilucoplan is in the interest of the participant in the investigator´s opinion
* Participant agrees to receive booster vaccinations against meningococcal infections during the study, if clinically indicated according to the local standard of care

Exclusion Criteria:

* Study participant met any mandatory investigational medicinal product (IMP) withdrawal or mandatory permanent discontinuation criteria in MG0014 or permanently discontinued IMP
* Participant has known positive serology for muscle-specific kinase
* Participant has known hypersensitivity to any components of the IMP
* Participant has a prior history of meningococcal disease

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2027-10-26 (Estimated); Study Completion 2027-11-19 (Estimated)

PRIMARY OUTCOMES:
Occurence of treatment emergent adverse events during the course of the study | Baseline (Day 1) to Safety Follow-up (up to Week 60)
  An adverse event (AE) is any untoward medical occurence in a patient or clinical investigation where the study participant administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Occurence of treatment-emergent serious adverse events (TESAEs) | Baseline (Day 1) to Safety Follow-up (up to Week 60)
  A serious adverse event (SAE) is defined as any untoward medical occurrence that, at any dose:
  Results in death Is life-threatening Requires inpatient hospitalization Results in persistent disability/incapacity Is a congenital anomaly/birth defect Important medical event.
Occurence of treatment-emergent advserse events leading to permanent withdrawal of investigational medicinal product | Baseline (Day 1) to Safety Follow-up (up to Week 60)
  An adverse event (AE) is any untoward medical occurence in a participant or clinical investigation administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. AEs leading to permanent withdrawal of study medication.
Occurence of treatment-emergent infections | Baseline (Day 1) to Safety Follow-up (up to Week 60)
  Percentage of participants who experienced treatment-emergent infections as adverse events.
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Plasma concentration of Zilucoplan at Week 52 | Week 52
  Blood samples for the measurement of plasma concentrations of Zilucoplan will be collected at Week 52.
Sheep red blood cell (sRBC) lysis activity at Week 52 | Week 52
  Blood samples for measurement of sRBC lysis will be collected at Week 52.
Blood complement component 5 (C5) levels at Week 52 | Week 52
  Blood samples for measurement of C5 will be collected at Week 52.
Myasthenia Gravis Activity of Daily Living (MG-ADL) score at Week 52 | Week 52
  The MG-ADL score is an 8-item patient-reported outcome (PRO) instrument. The MG-ADL targets symptoms and disability across ocular, bulbar, respiratory, and axial symptoms. The item responses are scored from 0 to 3, and the total score of MG-ADL is the sum of the 8 items and ranges from 0 to 24, with a higher score indicating more disability.
Quantitative Myasthenia Gravis (QMG) score at Week 52 | Week 52
  QMG score is a standardized and validated quantitative strength scoring system that was developed specifically for MG. The QMG total score is obtained by summing the responses to each individual item (13 items; Responses: None=0, Mild=1, Moderate=2, Severe=3). The score ranges from 0 to 39, with lower scores indicating lower disease activity.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (9):
- United States (2):
  - Mg0015 50168, Chicago, Illinois
  - Mg0015 50574, Denton, Texas
- Mg0015 40144, Milan, Italy
- Poland (2):
  - Mg0015 40774, Katowice
  - Mg0015 40218, Warsaw
- South Korea (2):
  - Mg0015 20104, Seoul
  - Mg0015 20220, Seoul
- United Kingdom (2):
  - Mg0015 40735, Glasgow
  - Mg0015 40736, London

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this study may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed.All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: https://www.Vivli.org